CLINICAL TRIAL: NCT05635552
Title: All Eyes on PCS - Analysis of the Retinal Microvasculature in Patients With Post-COVID-19 Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. Christoph Schmaderer, Principal Investigator, Technical University of Munich
Other Study IDs: 2022317PCS
Record Dates: First submitted 2022-11-18; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Long Covid19; Post COVID-19 Condition; Endothelial Dysfunction
Keywords: Retinal Vessel Analysis; Retinal microvasculature; Autoimmunity; Inflammation; Vasculopathy
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Autoimmune Diseases; Inflammation; Vascular Diseases | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva samples are collected from the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PCS patients: Patients with a COVID-19 infection at least 3 months ago (positive PCR or rapid antibody test) and PCS typical symptoms (e.g. fatigue, breast pain, heart palpitations, cognitive impairment) ongoing for at least 2 months and which cannot be explained by an alternative diagnosis.
  Interventions: Diagnostic Test: Dynamic retinal vessel analysis (DVA); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Biochemistry and immune phenotyping; Diagnostic Test: Handgrip strength test; Diagnostic Test: Questionnaires (Patient reported outcomes)
- COVID-19 recovered participants: Participants with Sars-CoV-2 infection at least 3 months ago (positive PCR or positive rapid antibody test) which are fully recovered.
  Interventions: Diagnostic Test: Dynamic retinal vessel analysis (DVA); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Biochemistry and immune phenotyping; Diagnostic Test: Handgrip strength test; Diagnostic Test: Questionnaires (Patient reported outcomes)
- COVID-19 infection naïve: No history of COVID-19 infection (exclusion via measurement of specific antibodies).
  Consists of an already established, pre-pandemic healthy cohort and a cohort recruited during the pandemic.
  Interventions: Diagnostic Test: Dynamic retinal vessel analysis (DVA); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Biochemistry and immune phenotyping

INTERVENTIONS:
Diagnostic Test: Dynamic retinal vessel analysis (DVA) — DVA is an established, non-invasive tool to measure the responsiveness of retinal vessels to flickering light. In addition static retinal vessel parameters are recorded.
Diagnostic Test: Optical coherence tomography (OCT) — OCT is an imaging technique which applies low-coherence light to capture high resolution images from the ocular fundus.
Diagnostic Test: Biochemistry and immune phenotyping — Blood sample collection for clinical chemistry and isolation of PBMCs for FACS analysis.
Diagnostic Test: Handgrip strength test — Measure the maximum isometric strength of the hand and forearm muscles and their fatiguability.
  Groups: COVID-19 recovered participants; PCS patients
Diagnostic Test: Questionnaires (Patient reported outcomes) — The questionnaires evaluate anxiety, depression, chronic fatigue, quality of life, and post-covid typical symptoms
  Groups: COVID-19 recovered participants; PCS patients

SUMMARY:
The goal of this observational, prospective study is to in depth analyze the retinal microvasculature in patients with Post-COVID-19 Syndrome (PCS). The main questions it aims to answer is:

Do patients with PCS show a prolonged endothelial dysfunction when compared with fully COVID-19 recovered participants? Does symptom severity in PCS patients correlate with the extend of endothelial dysfunction? Do these changes correlate with improvement in symptoms in the prospective observation?

DETAILED DESCRIPTION:
The investigators will recruit patients with PCS, fully COVID-19 recovered participants and COVID-19 infection naïve participants. After comprehensive clarification and given written informed consent, measurements will take place in the Klinikum rechts der Isar. To evaluate the retinal microvasculature dynamic retinal vessel analysis (DVA) and optical coherence tomography (OCT) are used. Patient reported outcomes (PROM) of PCS typical symptoms will be collected using standardized questionnaires. To ensure data quality the investigators will use standard operating procedures (SOP) for both technical measurements and data collection. For DVA measurements all examiners will be trained by a single experienced supervisor and must reach high image accuracy and quality in at least 10 volunteers. Examiners are only involved in data acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Post-COVID syndrome (positive PCR or positive rapid antibody test ≥3 months) with a currently existing, PCS-typical complaint complex, ongoing for at least 2 months and cannot be explained by an alternative diagnosis.
* Control group: recovered from COVID-19 infection (positive PCR or positive rapid antibody test ≥ 3 months) without residual symptoms.
* Healthy cohort: no history of COVID-19 infection

Exclusion Criteria:

* Missing or incomplete consent form
* Age < 18 years
* Pregnancy
* Malignancy
* Diseases associated with a significant change in life expectancy
* Autoimmune diseases of the rheumatological type
* Cataract
* Epilepsy
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample, Post-Covid ambulance, general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-02-21 (Estimated); Study Completion 2023-07-21 (Estimated)

PRIMARY OUTCOMES:
PCS patients show an impaired retinal vessel responsiveness when compared with fully recovered COVID-19 participants. | Baseline
  Static and dynamic parameters of the retinal vessel analysis.

SECONDARY OUTCOMES:
PCS patients show an impaired retinal vessel responsiveness at baseline when compared with infection naïve participants. | Baseline
  Static and dynamic parameters of the retinal vessel analysis.
PCS patients with improved symptoms show a change in retinal vessel responsiveness after 6 months when compared with baseline parameters. | Baseline to month 6
  Static and dynamic parameters of the retinal vessel analysis. Test items of the The COVID-19 Yorkshire Rehabilitation Scale (C19-YRS) and PCS questionnaire. Calculation of PCS severity scores (Bahmer, 2022) in each patient with a range of score values from zero (better outcome) to 59 (worse outcome). Comparison of retinal vessel parameters and PCS scores between Baseline and month 6.
Symptom severity of PCS in patients correlates with impaired retinal vessel responsiveness. | Baseline
  Correlation between PCS severity scores with static and dynamic parameters of the retinal vessel analysis.
PCS patients with impaired RVA analysis show elevated levels of markers of endothelial dysfunction and of chronic inflammation when compared with COVID-19 recovered cohort. | Baseline
  Measurement of markers of endothelial dysfunction:
  Concentration of: sICAM, sVCAM, Thrombomodulin, P-Selectin,E-Selectin, ADMA, SADMA, Endothelin-1, ACE-1, ACE-2, ANG-2, GDF-15.
  Measurement of markers of chronic inflammation Concentration of IFN-β, IFN-λ1,TNFa. Comparison of marker levels to the COVID-19 recovered cohort.
PCS patients with impaired RVA show a reactivation of EBV. | Baseline
  Using PCR to measure EBV reactivation in patients plasma .
Characterization of immune cell composition in PCS patients and comparison with COVID-19 recovered and COVID-19 infection naïve participants. | Baseline
  Using flow cytometry to detect different T-cell and monocyte subpopulations.
PCS patients show a decrease in vessel density in OCT-A when compared with COVID-19 recovered participants. | Baseline
  Parameters of OCT-A.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schmaderer, Prof. Dr., Principal Investigator — Technical University Munich
Locations (1):
- Klinikum rechts der Isar, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahmer T, Borzikowsky C, Lieb W, Horn A, Krist L, Fricke J, Scheibenbogen C, Rabe KF, Maetzler W, Maetzler C, Laudien M, Frank D, Ballhausen S, Hermes A, Miljukov O, Haeusler KG, Mokhtari NEE, Witzenrath M, Vehreschild JJ, Krefting D, Pape D, Montellano FA, Kohls M, Morbach C, Stork S, Reese JP, Keil T, Heuschmann P, Krawczak M, Schreiber S; NAPKON study group. Severity, predictors and clinical correlates of Post-COVID syndrome (PCS) in Germany: A prospective, multi-centre, population-based cohort study. EClinicalMedicine. 2022 Jul 18;51:101549. doi: 10.1016/j.eclinm.2022.101549. eCollection 2022 Sep. PMID 35875815
- [Derived] Kuchler T, Hausinger R, Braunisch MC, Gunthner R, Wicklein R, Knier B, Bleidissel N, Maier M, Ribero A, Lech M, Adorjan K, Stubbe H, Kotliar K, Heemann U, Schmaderer C. All eyes on PCS: analysis of the retinal microvasculature in patients with post-COVID syndrome-study protocol of a 1 year prospective case-control study. Eur Arch Psychiatry Clin Neurosci. 2024 Dec;274(8):1847-1856. doi: 10.1007/s00406-023-01724-5. Epub 2023 Dec 2. PMID 38041762
- [Derived] Kuchler T, Gunthner R, Ribeiro A, Hausinger R, Streese L, Wohnl A, Kesseler V, Negele J, Assali T, Carbajo-Lozoya J, Lech M, Schneider H, Adorjan K, Stubbe HC, Hanssen H, Kotliar K, Haller B, Heemann U, Schmaderer C. Persistent endothelial dysfunction in post-COVID-19 syndrome and its associations with symptom severity and chronic inflammation. Angiogenesis. 2023 Nov;26(4):547-563. doi: 10.1007/s10456-023-09885-6. Epub 2023 Jul 28. PMID 37507580